CLINICAL TRIAL: NCT06618001
Title: A Phase 1, First-in-Human, Dose Escalation Study of JNJ-89853413 for Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Neoplasms
Brief Title: A Study of JNJ-89853413 for Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 89853413AML1001; 89853413AML1001 (Other: Janssen Research & Development, LLC); 2024-513199-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Neoplasms
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-89853413 (Experimental): Participants will receive JNJ-89853413 in Part 1 (Dose escalation) of the study and the dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified. Participants in Part 2 (Dose expansion) will receive JNJ-89853413 at the RP2D determined in Part 1.
  Interventions: Drug: JNJ-89853413

INTERVENTIONS:
Drug: JNJ-89853413 — JNJ-89853413 will be administered.

SUMMARY:
The purpose of Part 1 (Dose Escalation) of the study is to assess the safety and tolerability, and to identify the recommended Phase 2 dose[s] (RP2D[s]) in participants with relapsed or refractory (R/R) acute myeloid leukemia (AML) (that is a type of blood cancer that has come back after treatment/or has stopped responding to treatment) or R/R higher-risk type of myelodysplastic neoplasms (MDS, type of blood cancer). The purpose of Part 2 (Cohort Expansion) is to further assess the safety, tolerability and efficacy in participants with R/R AML or higher-risk types of MDS.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis, per World Health Organization (WHO) 2022 criteria of:

  1. relapsed/refractory acute myeloid leukemia (AML)
  2. relapsed/refractory moderate high, high, or very high risk myelodysplastic neoplasms (MDS) per Molecular International Prognostic Scoring System (IPSS-M)
* Body weight greater than or equals to (>=) 40 kilograms (kg)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Have adequate renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Estimated Glomerular Filtration Rate (eGFR) >=40 milligrams per minute (mL/min)
* Participants must have laboratory parameters in the required range

Exclusion Criteria:

* Has a medical history of clinically significant pulmonary compromise, particularly the need for current supplemental oxygen use to maintain adequate oxygenation
* Has evidence of an uncontrolled systemic viral, bacterial, or fungal infection
* Has known allergies, hypersensitivity, or intolerance to the excipients of JNJ-89853413
* Had major surgery or had significant traumatic injury within 14 days of planned first dose of JNJ-89853413
* Has known active central nervous system involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-01-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AEs) by Severity | From screening untill 30 days after last dose of study drug (that is approximately 2.5 years)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLTs) | 14 days
  Participants with dose-limiting toxicity (DLT) will be assessed. DLT is defined as any toxicity that requires discontinuation of treatment, any Grade 5 toxicity; Non-hematologic Toxicity (Grade 3 or 4) and Hematologic Toxicity.

SECONDARY OUTCOMES:
Serum Concentration of JNJ- 89853413 | Approximately 2.5 years
  Serum samples will be analyzed to determine concentrations of JNJ-89853413 using a validated immunoassay method.
Area Under the Plasma Concentration-time (AUC[t]) Curve of JNJ-89853413 | Approximately 2.5 years
  AUC[t] is defined as the area under the plasma concentration time curve during a dosing interval at steady-state.
Maximum Serum Concentration (Cmax) of JNJ-89853413 | Approximately 2.5 years
  Cmax is defined as maximum serum concentration of JNJ-89853413.
Trough Observed Serum Concentration (Ctrough) of JNJ-89853413 | Approximately 2.5 years
  Ctrough is the trough observed serum concentration of JNJ-89853413.
Number of Participants with Presence of anti-drug Antibodies of JNJ-89853413 | Approximately 2.5 years
  Participants with anti JNJ-89853413 antibodies will be analyzed by a bridging electrochemiluminescence (ECL) enzyme linked immune assay.
Complete Response (CR) in Acute Myeloid Leukemia (AML) | Approximately 2.5 years
  CR is achieved when a participant has a best response of CR (complete response with partial hematologic recovery [CRh] or complete response with incomplete hematologic recovery [CRi]) according to the European Leukemia Network (ENL) 2022 criteria.
Overall Response (OR) in Myelodysplastic Neoplasms (MDS) | Approximately 2.5 years
  OR is achieved when a participant with MDS has a CR (any type, that is CRh or complete response with limited count recovery [CRL]), partial response (PR), or hematologic improvement (HI) according to the International Working Group (IWG) 2023 criteria.
Complete Response in MDS | Approximately 2.5 years
  CR is achieved when a participant has a best response of CR (including CRh/CRL) according to the IWG 2023 criteria.
Duration of Response (DOR) | Approximately 2.5 years
  DOR is defined for responsders only, as time from date of initial documentation of a response to the first documented evidence of no reponse, disease progression, relapse, initation of a new systemic anti-cancer therapy (besides hematopoietic stem cell transplant [HSCT]), or death, whichever comes first.
Time to response (TTR) | Approximately 2.5 years
  TTR is defined for responders only, as the time from the first dose of study drug to first qualifying response.
Number of Participants Achieving Transfusion independence | Approximately 2.5 years
  Transfusion independence is defined as the absence of red blood cell (RBC) and platelet transfusions for 8 weeks or longer after starting study treatment for participants with AML and 16 weeks or longer for participants with MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- Canada (3):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- Spain (3):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency